CLINICAL TRIAL: NCT00503685
Title: A Randomized Phase 2 Clinical Trial of IMC-A12, as a Single Agent or in Combination With Cetuximab, in Patients With Metastatic Colorectal Cancer With Disease Progression on Prior Anti-EGFR Therapy
Brief Title: Study Using IMC-A12 (Cixutumumab) With or Without Cetuximab in Participants With Metastatic Colorectal Cancer Who Have Failed a Treatment Regimen That Consisted of a Prior Anti-EGFR Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13936; CP02-0657 (Other: ImClone, LLC); CP13-0605 (Other: ImClone, LLC); I5A-IE-JAEL (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer
Keywords: Metastatic Colorectal Cancer with Disease Progression; Failed prior to Anti-EGFr Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — cixutumumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IMC-A12 (Experimental): Administered every 2 weeks
  Interventions: Biological: IMC-A12
- IMC-A12 + cetuximab (Experimental): Administered every 2 weeks
  Interventions: Biological: IMC-A12; Biological: cetuximab
- IMC-A12 + cetuximab [Kirsten rat sarcoma (K-ras) wild-type] (Experimental): Participants who have experienced confirmed partial response (PR) or stable disease (SD) ≥ 24 weeks on a prior anti-EGFR-containing therapy followed by disease progression are enrolled in this arm.
  Interventions: Biological: IMC-A12; Biological: cetuximab

INTERVENTIONS:
Biological: IMC-A12 — 10 milligrams/kilogram (mg/kg) intravenous infusion every 2 weeks.
  Other Names: Cixutumumab; LY3012217
Biological: cetuximab — Participants will receive cetuximab 500 milligrams/square meter (mg/m²) intravenous over 2 hours every 2 weeks.
  Other Names: Erbitux®
  Arms: IMC-A12 + cetuximab; IMC-A12 + cetuximab [Kirsten rat sarcoma (K-ras) wild-type]

SUMMARY:
Participants with metastatic Colorectal Cancer (mCRC) who have progressed on a prior Anti-epidermal growth factor receptor (EGFR) regimen randomized to receive IMC-A12 monotherapy or combination therapy with cetuximab to assess response, survival, durations of response, safety and tolerability as well as pharmacodynamics of IMC-A12 and cetuximab

ELIGIBILITY:
Inclusion Criteria

* The participant has histologically or cytologically-confirmed colorectal cancer with metastatic disease documented on diagnostic imaging studies
* The participant has measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded), measuring ≥ 2 centimeter (cm) on conventional measurement techniques or ≥ 1 cm on spiral computed tomography (CT) scan
* The participant has clinical documentation of disease progression during treatment or within 6 weeks after receiving the last dose of a therapeutic regimen for metastatic disease containing an anti-EGFR-component (cetuximab or panitumumab). Toxicity or planned treatment break will not be regarded as adequate evidence of disease progression and such participants will not be eligible for this trial
* The participant has received at least one prior standard and/or investigational regimen for metastatic disease
* The participant is age ≥ 18 years
* The participant has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1 (Karnofsky ≥ 80%
* The participant has adequate hematologic function as defined by an absolute neutrophil count ≥ 1500/microliter (μL), hemoglobin ≥ 9 grams/deciliter (g/dL), and a platelet count ≥ 100,000/μL
* The participant has adequate hepatic function as defined by a total bilirubin ≤ 1.5 x the upper limit of normal (ULN), and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x the ULN (or ≤ 5 x the ULN in the presence of known liver metastases)
* The participant has adequate coagulation function as defined by international normalized ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) ≤ 1.5 x the ULN. Participants on full-dose anticoagulation must be on a stable dose of oral anticoagulant or low molecular weight heparin, and if on warfarin must have an INR between 2 and 3 and have no active bleeding or pathological condition that carries a high risk of bleeding (for example, tumor involving major vessels or invading the rectal lumen, or known varices)
* The participant has adequate renal function as defined by serum creatinine ≤ 1.5 x the institutional ULN or creatinine clearance ≥ 60 milliliters/minute (mL/min) for participants with creatinine levels above the ULN, as well as urine protein ≤ 1+ on urine dipstick or routine urinalysis [(UA), if urine dipstick/routine UA indicates ≥ 2+ protein, a 24-hour urine collection for protein must demonstrate < 1000 milligrams (mg) of protein in 24 hours to allow participation in the study]
* The participant has fasting serum glucose < 120 milligrams/deciliter (mg/dL) or below the ULN
* The participant has a life expectancy of > 3 months
* Because the teratogenicity of IMC-A12 (cixutumumab) is not known, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* The participant has the ability to understand and the willingness to sign a written informed consent document
* The participant has a tumor that is K-ras wild-type (absence of mutations at codon 12 or 13, as determined by the DxS K-ras Mutation Kit [polymerase chain reaction (PCR)-based analysis]).
* The participant experienced either a confirmed partial response or stable disease of ≥ 24 weeks duration during prior treatment with a cetuximab- or panitumumab-containing regimen except for participants with uridine diphosphate glucuronosyltransferase 1A1 (UGT1A1) promoter polymorphism, for example, Gilbert syndrome, confirmed by genotyping or Invader®UGT1A1 Molecular Assay prior to enrollment. Participants enrolled with Gilbert Syndrome must have a total bilirubin ≤ 3 x ULN. If the participant has liver metastases, total bilirubin must be ≤ 3 x ULN.

Exclusion Criteria

* The participant has received chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or has not recovered from adverse events due to agents administered more than 4 weeks earlier. Neurotoxicity, if present, must have recovered to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version 3.0 grade ≤ 2.
* The participant is receiving any other investigational agent(s).
* The participant has a history of treatment with other agents targeting the insulin-like growth factor receptor (IGFR).
* The participant has known brain or leptomeningeal metastases.
* The participant has a history of primary central nervous system tumors, seizures not well controlled with standard medical therapy, or history of stroke within 6 months prior to randomization.
* The participant has a history of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab or IMC-A12 (cixutumumab).
* The participant has poorly controlled diabetes mellitus. Participants with a history of diabetes mellitus are allowed to participate, provided that their blood glucose is within normal range (fasting glucose < 120 mg/dL or below ULN) and that they are on a stable dietary or therapeutic regimen for this condition.
* The participant has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, uncontrolled hypertension, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* The participant is pregnant or lactating.
* The participant is known to be positive for infection with the human immunodeficiency virus.
* The participant is receiving therapy with immune modulators such as cyclosporine or tacrolimus.
* The participant has a history of another primary cancer, with the exception of: a) curatively resected nonmelanomatous skin cancer; b) curatively treated cervical carcinoma in-situ; or c) other primary solid tumor curatively resected treated with no known active disease present and no treatment administered for the last 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (4):
- United States (4):
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, New Haven, Connecticut
  - ImClone Investigational Site, Buffalo, New York
  - ImClone Investigational Site, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with progressive disease (PD) or death are considered having completed study.
Groups:
- IMC-A12: Participants received 10 milligrams/kilogram (mg/kg) IMC-A12 intravenous infusion over 1 hour every 2 weeks until there was evidence of PD, unacceptable toxicity, or withdrawal of consent.
- IMC-A12 + Cetuximab: Participants received cetuximab 500 milligrams/square meter (mg/m²) intravenous infusion over 2 hours followed by 10 mg/kg IMC-A12 intravenous infusion over 1 hour. This sequence was repeated every 2 weeks until there was evidence of PD, unacceptable toxicity, or withdrawal of consent.
- IMC-A12 + Cetuximab (K-ras Wild-type): Participants with Kirsten rat sarcoma (K-ras) wild-type who experienced confirmed partial response (PR) or stable disease (SD) ≥ 24 weeks on a prior anti-epidermal growth factor receptor (EGFR)-containing therapy followed by disease progression were enrolled in this arm.
  Participants received cetuximab 500 mg/m² intravenous infusion over 2 hours followed by 10 mg/kg IMC-A12 intravenous infusion over 1 hour. This sequence was repeated every 2 weeks until there was evidence of PD, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Started | 23 | 22 | 20
Received at Least 1 Dose of Study Drug | 23 | 21 | 20
Completed | 23 | 19 | 18
Not Completed | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Eligibility Criteria Not Met | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized/enrolled participants who received at least 1 dose of study drug.
Groups:
- IMC-A12: Participants received 10 mg/kg IMC-A12 intravenous infusion over 1 hour every 2 weeks until there was evidence of PD, unacceptable toxicity, or withdrawal of consent.
- IMC-A12 + Cetuximab: Participants received cetuximab 500 mg/m² intravenous infusion over 2 hours followed by 10 mg/kg IMC-A12 intravenous infusion over 1 hour. This sequence was repeated every 2 weeks until there was evidence of PD, unacceptable toxicity, or withdrawal of consent.
- IMC-A12 + Cetuximab (K-ras Wild-type): Participants with K-ras wild-type who experienced confirmed PR or SD ≥ 24 weeks on a prior anti-EGFR-containing therapy followed by disease progression were enrolled in this arm.
  Participants received cetuximab 500 mg/m² intravenous infusion over 2 hours followed by 10 mg/kg IMC-A12 intravenous infusion over 1 hour. This sequence was repeated every 2 weeks until there was evidence of PD, unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type) | Total
Number analyzed (Participants) | 23 | 21 | 20 | 64
Age, Continuous [Median (Full Range); unit: years] | 59.3 (8.94) [41 to 79] | 62.6 (12.40) [40 to 84] | 61.7 (7.89) [44 to 70] | 60.5 (9.84) [40 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 10 | 33
  Male | 9 | 12 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 7
  Not Hispanic or Latino | 21 | 18 | 18 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 17 | 17 | 51
  Black | 4 | 2 | 2 | 8
  Asian | 1 | 1 | 1 | 3
  Hispanic | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 21 | 20 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response [PR, Objective Response Rate (ORR)]
Description: ORR is the percentage of participants with a confirmed CR or PR, as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. CR is the disappearance of all target and non-target lesions; PR is a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesions. ORR is calculated as a total number of participants with CR or PR from start of the treatment until disease progression or recurrence divided by the total number of participants treated, then multiplied by 100.
Time Frame: Start of randomization/treatment to date of objective progressive disease (PD) up to 28.3 weeks
Population: All randomized/enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 23 | 21 | 20
percentage of participants | 0.0 [0.0 to 14.8] | 4.8 [0.1 to 23.8] | 0.0 [0.0 to 16.8]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the duration from the date of randomization/treatment to the date of PD or death from any cause. PD was determined using RECIST criteria version 1.0. PD is ≥20% increase in sum of longest diameter of target lesions or the appearance of new lesions. Participants who had no PD or death at the time of the data inclusion cutoff, PFS was censored at their last tumor assessment prior to the cutoff date. Participants who began a new antitumor treatment before evidence of PD were categorized as PD.
Time Frame: Randomization/treatment to measured PD up to 28.3 weeks
Population: All randomized/enrolled participants who received at least 1 dose of study drug. The number of participants censored was 0 for IMC-A12 group, 1 for IMC-A12 + cetuximab group and 1 for IMC-A12 + cetuximab (K-ras wild-type) group.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 23 | 21 | 20
weeks | 5.9 [5.6 to 5.9] | 6.1 [5.6 to 6.4] | 9.4 [5.6 to 11.6]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration from the date of randomization/treatment to the date of death from any cause. Participants who were alive at the time of the data inclusion cutoff, OS was censored at the last date the participant was known to be alive.
Time Frame: Randomization/treatment to date of death from any cause up to 26.9 months
Population: All randomized/enrolled participants who received at least 1 dose of study drug. The number of participants censored was 5 for IMC-A12 group, 4 for IMC-A12 + cetuximab group and 11 for IMC-A12 + cetuximab (K-ras wild-type) group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 23 | 21 | 20
months | 5.7 [3.4 to 7.9] | 4.5 [2.8 to 13.3] | 10.9 [5.5 to NA] — Upper limit of 95% confidence interval was not estimable due to high censoring rate.

4. Secondary Outcome: Duration of Stable Disease (SD)
Description: The duration of SD is measured from the date of randomization/treatment until the date of PD. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. RECIST criteria version 1.0 was used to asses PR and PD. PR is ≥30% decrease in sum of longest diameter of target lesions. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion. Participants who had no PD or death at the time of the data inclusion cutoff, duration of SD was censored at their last tumor assessment prior to the cutoff date.
Time Frame: Time from randomization/treatment to first date of PD up to 28.3 weeks
Population: All randomized/enrolled participants who received at least 1 dose of the study drug and achieved SD or better. The number of participants censored was 0 for IMC-A12 group, 0 for IMC-A12 + cetuximab group and 1 for IMC-A12 + cetuximab (K-ras wild-type) group.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 3 | 3 | 12
weeks | 11.1 [10.7 to 12.3] | 15.4 [11.4 to 28.3] | 11.6 [9.0 to 17.9]

5. Secondary Outcome: Duration of Overall Response
Description: The duration of overall response (CR or PR) was defined as the time from first objective status assessment of CR or PR to the first time of PD or death due to any cause. CR, PR and PD were determined using RECIST criteria version 1.0. CR is the disappearance of all target and non-target lesions; PR is a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesions; PD is ≥20% increase in sum of longest diameter of target lesions or the appearance of new lesions. For participants with CR or PR who had no PD or death at the time of the data inclusion cutoff, the duration of overall response was censored at their last tumor assessment prior to the cutoff date. Duration of overall response was not analyzed due to low number of participants with CR or PR.
Time Frame: Time of response to time of measured PD or death up to 161 days
Population: Zero participants analyzed. Duration of Response for CR or PR data was not collected for analysis due to N=0 CR and N=1 PR.
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs)
Description: Data presented are the number of participants who experienced nonserious adverse events (AEs) during the study including the 30-day follow-up. A summary of serious AEs (SAEs) and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Randomization/treatment up to 26.9 months
Population: All randomized/enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 23 | 21 | 20
Participants | 18 | 19 | 20

7. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Severe Adverse Events
Description: Data presented are the number of participants who experienced serious adverse events (SAEs) or death during the study including the 30-day follow-up. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Randomization/treatment up to 26.9 months
Population: All randomized/enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 23 | 21 | 20
Participants
  SAEs | 7 | 6 | 4
  Death Due to PD | 1 | 0 | 0
  Death Due to SAE | 0 | 1 | 0

8. Secondary Outcome: Maximum Concentration (Cmax)
Time Frame: Week 1 (Initial dose), Week 3 (Dose 2), Week 5 (Dose 3), Week 7 (Dose 4), Week 9 (Dose 5), and Week 11 (Dose 6)
Population: Zero participants analyzed. PK data was not collected for analysis due to the low number of participants in PK.
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Minimum Concentration (Cmin)
Time Frame: Week 1 (Initial dose), Week 3 (Dose 2), Week 5 (Dose 3), Week 7 (Dose 4), Week 9 (Dose 5), and Week 11 (Dose 6)
Population: Zero participants analyzed. PK data was not collected for analysis due to the low number of participants in PK.
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Area Under Serum Concentration (AUC)
Time Frame: Week 1 (Initial dose), Week 3 (Dose 2), Week 5 (Dose 3), Week 7 (Dose 4), Week 9 (Dose 5), and Week 11 (Dose 6)
Population: Zero participants analyzed. PK data was not collected for analysis due to the low number of participants in PK.
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR, Response Rate) in Participants With Kirsten Rat Sarcoma (K-ras) Mutations
Description: The response rate in participants with K-ras mutations was not collected for analysis.
Time Frame: Treatment up to 26.9 months
Population: Zero participants analyzed. Response rate data was not collected for analysis due to N=0 CR and N=1 PR.
Arm/Group | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 0

12. Secondary Outcome: Expression of Type I Insulin-Like Growth Factor Receptors (IGF-IR)
Time Frame: Randomization/treatment up to 26.9 months
Population: Zero participants analyzed. No data collected for analysis.
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Expression of IGF Binding Proteins (IGFBP2, IGFBP3)
Time Frame: Randomization/treatment up to 26.9 months
Population: Zero participants analyzed. No data collected for analysis.
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | IMC-A12 | IMC-A12 + Cetuximab | IMC-A12 + Cetuximab (K-ras Wild-type)
Serious Adverse Events (participants affected / at risk) | 7/23 | 6/21 | 4/20
Other Adverse Events (participants affected / at risk) | 18/23 | 19/21 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 (N=23) | IMC-A12 + Cetuximab (N=21) | IMC-A12 + Cetuximab (K-ras Wild-type) (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Disease progression (General disorders) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 (N=23) | IMC-A12 + Cetuximab (N=21) | IMC-A12 + Cetuximab (K-ras Wild-type) (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (6) | 4 (5)
Nausea (Gastrointestinal disorders) | 3 (4) | 6 (9) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (3) | 3 (5) | 4 (4)
Fatigue (General disorders) | 7 (9) | 8 (11) | 8 (9)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (2) | 2 (3)
Blood bilirubin increased (Investigations) | 2 (3) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 4 (5) | 2 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 3 (5) | 5 (7)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (10) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (4) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (4) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (19) | 9 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 7 (7)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 6 (7)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.